CLINICAL TRIAL: NCT03061448
Title: Internet-based Exposure Therapy for Panic Disorder: A Randomized Controlled Pilot Study
Brief Title: Internet-based Exposure Therapy for Panic Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Erik Andersson, PhD, psychologist, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016/2422-31
Record Dates: First submitted 2017-02-19; First posted 2017-02-23 (Actual); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Panic Disorder With Agoraphobia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inhibitory learning based treatment (Experimental): The experimental group will go through Internet-based treatment. The exposure treatment is 8 weeks long and based on the principles of inhibitory learning, i.e. the participant is instructed to stay in the frightening situation until his/her expectancy has been maximally violated.
  Interventions: Behavioral: Internet-based cognitive-behavior therapy
- Habituation based treatment (Active Comparator): The active comparator group will also go through Internet-based treatment. The exposure treatment is 8 weeks long and based on the principles of emotional processing theory, i.e. the participant is instructed to stay in the frightening situation until anxiety has declined (habituated).
  Interventions: Behavioral: Internet-based cognitive-behavior therapy

INTERVENTIONS:
Behavioral: Internet-based cognitive-behavior therapy — Internet-based cognitive-behavior therapy on a safe internet platform. Treatment is divided into eight modules, each containing homework assignments . The participants will be assigned a therapist that they can contact through a message system in the platform and expect answer within 24 hours.

SUMMARY:
The purpose of this study is examine if an internet-based exposure therapy based on inhibitory learning is feasible, acceptable and effective in reducing panic symptoms amongst patients who suffer from panic disorder and agoraphobia.

DETAILED DESCRIPTION:
Trial objectives: Primary objective is to examine if an internet-based exposure therapy based on inhibitory learning is effective in reducing panic symptoms. The secondary objective is to study if the protocol is feasible and acceptable. Secondary objective is measured is examined on 1) number of participants completing the study protocol, 2) participants' satisfaction with the treatment, 3) therapists' ratings of acceptability. The aim of this study is to assess the feasibility, and pilot the design and delivery of a RCT that will subsequently form the framework for a larger RCT to evaluate the effectiveness of an exposure protocol based on inhibitory learning.

Trial Design: Randomized controlled pilot study with two groups randomly assigned to either Internet-based exposure therapy based on the principles of inhibitory learning or Internet-based exposure therapy based on the principles of habituation Duration: Eight weeks Primary Endpoint: Change in panic symptoms from baseline to Week 8. Efficacy Parameters: Panic Disorder Severity Scale - Self rated (PDSS-SR) Safety Parameters: Adverse Events is assessed weekly via the internet. Description of Trial Subjects: Patients > 18 years old with a PDSS-SR score more than 6 points Number of Subjects: 80

ELIGIBILITY:
Inclusion Criteria:

* Outpatients
* ≥ 18 years
* Situated in Sweden
* Informed consent
* Panic Disorder Severity Scale - self rated score more than 6 points

Exclusion Criteria:

* Substance dependence during the last six months
* Post traumatic stress disorder, bipolar disorder or psychosis
* Symptoms better explained by axis 2 diagnosis (e.g. autism or borderline personality disorder)
* MADRS-S score above 25 points
* Psychotropic medication changes within one months prior to treatment that could affect target symptoms.
* Received exposure based Cognitive behavior therapy (CBT) for pathological worry the last 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Panic Disorder Severity Scale - Self rated (PDSS-SR) | Week 0, Week 8
  Change in panic symptoms from baseline to Week 8

SECONDARY OUTCOMES:
Credibility/Expectancy Questionnaire (CEQ) | Week 2
  Measuring treatment expectancy and rationale credibility for use in clinical outcome studies
Client Satisfaction Questionnaire (CSQ) | Week 8
  To assess client satisfaction with treatment
Adverse events scale | Week 8
  To assess any adverse events caused by the treatment
Patient Health Questionnaire (PHQ-9) | Week 0, Week 8
  Change in depression from baseline to Week 8
Anxiety Sensitivity Index (ASI) | Week 0, Week 8
  Change in fear of anxiety-related physical sensations
Agoraphobic Cognitions Questionnaire (ACQ) | Week 0, Week 8
  Change in fear of fear in agoraphobics
Body Sensations Questionnaire (BSQ) | Week 0, Week 8
  Change in fear of bodily sensations in agoraphobics
Brunnsviken Quality of Life Questionnaire (BBQ) | Week 0, Week 8
  Change in self-perceived quality of life from baseline to week 8
WHO Disability Assessment Schedule 2.0 (WHODAS 2.0) | Week 0, Week 8
  Change in functioning and disability
Generalised Anxiety Disorder Assessment (GAD-7) | Week 0, Week 8
  Screening tool and severity measure for generalised anxiety disorder
The Cardiac Anxiety Questionnaire (CAQ) | Week 0, Week 8
  Change in heart-focused anxiety from baseline to week 8
HA-NI-SSD Symptom Preoccupation Scale - testversion (SPSt) | Week 0, Week 8
  Change in preoccupation of symptoms from baseline to week 8

CONTACTS AND LOCATIONS:
Overall Officials: Erik M Andersson, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Sweden